CLINICAL TRIAL: NCT01794091
Title: Comprehensive Stress-Perfusion Cardiac MRI Assessment of Diabetic Cardiomyopathy: Prognostic Role of the Fibrotic Index
Brief Title: Detection of Diffuse Scar in Patients With Diabetes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants were enrolled in the trial.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Raymond Y. Kwong, MD, Associate Professor - Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: Fibrotic Index in Diabetics
Record Dates: First submitted 2013-02-15; First posted 2013-02-18 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type II
Keywords: Cardiac Magnetic Resonance Imaging; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eplerenone (Experimental): In a subgroup of 50 patients, 25 will be randomized to eplerenone to assess effects on fibrotic index pre- and post-6 months of therapy.
  Interventions: Drug: Eplerenone
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplerenone — Eplerenone 25 mg daily for 6 months
  Arms: Eplerenone
Drug: Placebo
  Arms: Sugar pill

SUMMARY:
People with diabetes are at an increased risk of heart attacks and heart failure, and it is important to be able to treat people with diabetes who are at risk for heart disease to prevent these outcomes. This study is looking at the importance of "diffuse scar tissue" that is found in the heart of diabetic people. We have discovered a way to detect diffuse scar tissue by cardiac MRI, a non-invasive test. In this study, we do cardiac MRI on diabetics with low risk stress test results and follow them for 5 years to see if the measure of scar tissue in the heart by MRI is related to events. If this study is positive, we will be able to use cardiac MRI scar tissue measurements to target those patients with diabetes who are at highest risk.

DETAILED DESCRIPTION:
This study will be conducted in TWO (2) PHASES:

Phase 1: Prospective cohort study of patients with diabetes mellitus, in which index cardiac MRI will be done after screening to determine FIBROTIC INDEX. Patients are subsequently followed for 5 years for a primary endpoint (composite cardiovascular event).

Phase 2: Of the patients with "HIGH" FIBROTIC INDEX, 50 patients will be randomly selected and randomized 1:1 to placebo:eplerenone 25 mg daily for 6 months, and a repeat cardiac MRI will be done to assess the fibrotic index post-treatment.

Phase 2 is a PILOT study of 50 patients.

The inclusion/exclusion criteria for the different phases is shown below.

ELIGIBILITY:
For PHASE I (Prospective Cohort Study to determine prognostic value of fibrotic index)

Inclusion Criteria:

* Diabetes mellitus, type II
* Age >= 40 years
* UKPDS 10 year Risk Score > 15%
* Low risk stress test (defined explicitily in our protocol)

Exclusion Criteria:

* suspected or confirmed myocarditis or infiltrative disease (including hemochromatosis, sarcoid, or amyloid)
* history of prior MI or coronary revascularization (by Q waves on electrocardiogram in 2 contiguous leads or by clinical history)
* clinical HF (with prior hospital admission for HF or documentation of reduced LV ejection fraction after index CMR)
* metallic hazards
* hematocrit < 30% (within 1 year of nuclear stress test) or history of active bleeding (within 3 months of stress test)
* estimated GFR (by Modified Diet in Renal Disease) < 45 ml/min/1.73m2 (within 2 weeks of planned CMR)
* pregnancy
* severe non-cardiac illness that or prognosis (e.g., end stage liver disease, malignancy, advanced HIV/AIDS)

For PHASE 2:

Inclusion Criteria:

* Included in Phase I
* Systolic blood pressure > 140 mmHg on two occasions (at the initial nuclear stress test and at the index cardiac MRI)

Exclusion criteria:

1. Concomitant cytochrome P450 (CYP3A4) inhibitors or inducers;
2. Concomitant potassium supplementation or potassium sparing diuretics;
3. Concomitant use of both ACE inhibitor and ARB therapy (at any dose);
4. Renal dysfunction (GFR < 50 ml/min or serum creatinine > 1.5 mg/dL (as assessed at time of index CMR);
5. Any urine microalbuminuria (as assessed at time of index CMR);
6. Baseline (pre-therapy) serum potassium > 5.0 mEq/L;
7. Lack of reliable telephone contact number for relaying results or the need to discontinue drug therapy;
8. Age > 75 years (given the tendency toward renal insufficiency not captured by GFR, dehydration and/or concomitant illness)
9. Women able to become pregnant (given the undefined risk of eplerenone therapy in pregnant women and newborns).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
All cause mortality, cardiovascular death, myocardial infarction or stroke | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States